CLINICAL TRIAL: NCT06220760
Title: Outcomes of Placenta Accreta Spectrum Disorders Surgery in Relation to Placenta Accreta Scoring Index
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Nagy Zaki, Clinical professor, Assiut University
Other Study IDs: US in Placenta accreta
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Placenta Previa; Placenta Accreta
MeSH Terms: conditions — Placenta Previa; Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — The use of US to calculate placenta accreta index

SUMMARY:
Using of Ultra sound in assessment of Placenta Accreta Index to predict the surgical outcomes of Placenta accreta

DETAILED DESCRIPTION:
Placenta accreta is a substantially life-threatening condition and one of the causes of maternal morbidity and mortality in the world. According to study done in United Kingdom, The estimated incidence of placenta accreta/increta/percreta was 1.7 per 10,000 maternities overall and 577 per 10,000 in women with both a previous caesarean delivery and placenta previa [1]. in a tertiary south Italian center, The incidence increased from 0.12% during the 1970s, to 0.31% during the 2000s [2].While in USA, the prevalence of placenta accreta was 3.7 per 1000 deliveries [3].

This increase is due to many factors. A scar of previous uterine surgery is a major risk factor for placenta accreta. Caesarean section scar is the most common one of uterine scars according to [4] especially in presence of placenta previa where the risk of placenta accreta was 3%, 11%, 40%, 61%, and 67% for the first, second, third, fourth, and fifth or greater repeat cesarean deliveries, respectively. [5] reported that both cesarean delivery morbidity and placenta accreta were positively associated with age >30 years. Previous myomectomy, multi parity, vigorous curettage are other risk factors as said [6]. More ever sub mucous leiomyoma and thermal ablation are also contributing factors to Placenta accreta [7] and lastly [8] said that uterine artery embolization is considered as a risk factor for occurrence of placenta accreta. Contrarily, inter pregnancy interval more than 60 months was associated with decreased risk of placenta accreta [9].

Because placenta accreta can lead to life-threatening blood loss, identification of these high-risk patients would be helpful in management of the pregnancy in addition to enabling the surgeon to be prepared adequately before the time of delivery. Many studies have been done on identification of placenta accreta in the third trimester by 2D ultrasound and color Doppler. There are many modalities for detection of placenta accreta ante natally [10] used 2D ultrasound and color doppler for detection of placenta accreta in 3rd trimester with sensitivity and specificity; 95.24% and 94.74% respectively for ultrasound with the most prominent feature presence of multiple lakes that represented dilated vessels extending from the placenta through the myometrium. For Doppler, the most prominent feature was the presence of interphase hypervascularity with abnormal vessels linking the placenta to the bladder, and the rate was 95.24%.

As for surgery for placenta accreta, planned caesarean hysterectomy is recommended to reduce mortality and morbidity, but fertility is lost. Antenatal diagnosis of placenta accreta spectrum (PAS) can ensure multidisciplinary management at center of excellence which can reduce maternal and fetal complications. This can be established by a scoring system which provides a standardized criterion for the diagnosis and management Placenta Accreta Index (PAI).

Instead of adhering to the conventional approach that involves an elective caesarean hysterectomy based on antenatal imaging, more suitable approaches should be considered from the spectrum of hemostatic and fertility-preserving options available. In our study we will investigate if the degree of adherence is related to the PAI score. Therefore, we can predict cases which will need conservative surgery or peripartum hysterectomy. And so that the surgeon be preplanned to do either hysterectomy or conservative surgery

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women with gestational age 32 weeks or more
2. singleton pregnancy
3. known to have placenta previa (lower edge of the placenta within 5 cm from internal Os )
4. with at least previous 1 cesarean section

Exclusion Criteria:

1. the patient is active in labor
2. haemodynamically unstable

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with Previous Scar of cesarean section who are 32weeks of gestation or more who are known to be Placenta previa
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
to decide If placenta accreta index (PAI) can predict suitable type of operation needed whether Conservative management/fertility-sparing techniques or Caesarean hysterectomy | 23 months

SECONDARY OUTCOMES:
Incidence of fetal complication associated with placenta accreta | 23 months
Incidence of maternal complications associated with placenta accreta | 23 months
The need for ICU admission after placenta accreta surgery and its duration | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Nagy, MD, Study Chair — Assiut University; Mansour Khalifa, MD, Study Director — Assiut University; Mostafa Hussien, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23300807/